CLINICAL TRIAL: NCT00572845
Title: Energy Costs of Spasticity in Spinal Cord Injury: A Pilot Investigation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit enough participants.
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: HM11352
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Basal Energy Expenditure; Spasticity
Keywords: Basal Energy Expenditure; Spasticity; Modified Ashworth Scale; Penn Spasm Frequency Score
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Weaning of Spasticity Medication over a three day period while measuring Modified Ashworth Scale and Penn Spasm Frequency Score. Then titration of medication back to previous dose over a three day period.
  Interventions: Other: Weaning of Antispasticity Medication

INTERVENTIONS:
Other: Weaning of Antispasticity Medication — Weaning of antispasticity medication over a three day period and then titration back to previous dose over a three day period.

SUMMARY:
The purpose of this study is to determine if there is a relationship between spasticity and relative changes in Basal Energy Expenditure in persons with spinal cord injury.

DETAILED DESCRIPTION:
Obesity is at epidemic proportions in the population with spinal cord injury (SCI), and is likely the mediator of the metabolic syndrome in this special population. Recent literature reviews have suggested that obesity is present in > 67% of persons with SCI. Additionally, recent studies have demonstrated the causal relationship between adipose tissue accumulation and vascular inflammation, dyslipidemia, insulin resistance / glucose intolerance, hypertension and thromboemboli.

Obesity in SCI occurs because of acute and ongoing positive energy balance, i.e., greater caloric intake than energy expenditure. Total Daily Energy Expenditure (TDEE) in SCI is reduced primarily because of muscular atrophy and diminished muscular contraction; pharmacological treatment of spasticity possibly reduces energy expenditure (EE) even further, but has not been evaluated to date. TDEE is comprised of three components: Basal Energy Expenditure (BEE), Thermic Effect of Activity (TEA) and Thermic Effect of Food (TEF). Of the three, BEE contributes the greatest amount (65-75% TDEE) and is the most sensitive to changes in spasticity.

Dampening spasticity has been reported to increase weight gain and necessitate reduced caloric intake in a child with spastic quadriplegia. Similarly, athetosis in patients with cerebral palsy increased resting metabolic rate (RMR) as compared to control subjects with no athetotic movements. Although several studies have reported energy requirements for persons with neurodevelopmental disabilities, and even SCI, however, none have attempted to measure the metabolic effect of spasticity.

ELIGIBILITY:
Inclusion Criteria:

* C1-T10 SCI at least 1 year post injury
* Spasticity in the legs
* Veteran

Exclusion Criteria:

* Recent increase in spasticity
* Botox within 6 months
* Phenol within 2 years
* Prior surgery for spasticity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Increase in Basal Energy Expenditure | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: David R Gater, MD, PhD, Principal Investigator — McGuire VA Medical Center; David X Cifu, MD, Study Chair — VCU Department of Physical Medicine and Rehabilitation
Locations (1):
- McGuire VA Medical Center, Richmond, Virginia, United States

REFERENCES:
- [Background] Buchholz AC, McGillivray CF, Pencharz PB. Differences in resting metabolic rate between paraplegic and able-bodied subjects are explained by differences in body composition. Am J Clin Nutr. 2003 Feb;77(2):371-8. doi: 10.1093/ajcn/77.2.371. PMID 12540396
- [Background] Gater DR Jr. Obesity after spinal cord injury. Phys Med Rehabil Clin N Am. 2007 May;18(2):333-51, vii. doi: 10.1016/j.pmr.2007.03.004. PMID 17543776
- [Background] Bauman WA, Spungen AM, Wang J, Pierson RN Jr. The relationship between energy expenditure and lean tissue in monozygotic twins discordant for spinal cord injury. J Rehabil Res Dev. 2004 Jan-Feb;41(1):1-8. doi: 10.1682/jrrd.2004.01.0001. PMID 15273892
- [Background] Hemingway C, McGrogan J, Freeman JM. Energy requirements of spasticity. Dev Med Child Neurol. 2001 Apr;43(4):277-8. doi: 10.1017/s0012162201000524. PMID 11305407
- [Background] Dickerson RN, Brown RO, Gervasio JG, Hak EB, Hak LJ, Williams JE. Measured energy expenditure of tube-fed patients with severe neurodevelopmental disabilities. J Am Coll Nutr. 1999 Feb;18(1):61-8. doi: 10.1080/07315724.1999.10718828. PMID 10067660
- [Background] Cox SA, Weiss SM, Posuniak EA, Worthington P, Prioleau M, Heffley G. Energy expenditure after spinal cord injury: an evaluation of stable rehabilitating patients. J Trauma. 1985 May;25(5):419-23. PMID 3999162
- [Background] Rodriguez DJ, Benzel EC, Clevenger FW. The metabolic response to spinal cord injury. Spinal Cord. 1997 Sep;35(9):599-604. doi: 10.1038/sj.sc.3100439. PMID 9300966
- [Background] Rodriguez DJ, Clevenger FW, Osler TM, Demarest GB, Fry DE. Obligatory negative nitrogen balance following spinal cord injury. JPEN J Parenter Enteral Nutr. 1991 May-Jun;15(3):319-22. doi: 10.1177/0148607191015003319. PMID 1907682
- [Background] Bohannon RW, Smith MB. Interrater reliability of a modified Ashworth scale of muscle spasticity. Phys Ther. 1987 Feb;67(2):206-7. doi: 10.1093/ptj/67.2.206. PMID 3809245
- [Background] Penn RD. Intrathecal baclofen for severe spasticity. Ann N Y Acad Sci. 1988;531:157-66. doi: 10.1111/j.1749-6632.1988.tb31822.x. No abstract available. PMID 3382141
- [Background] Gorgey AS, Gater DR Jr. Prevalence of Obesity After Spinal Cord Injury. Top Spinal Cord Inj Rehabil. 2007 Spring;12(4):1-7. doi: 10.1310/sci1204-1. PMID 29472754